CLINICAL TRIAL: NCT01440049
Title: Assessment Of Follow-Up Methods For Patients Treated In The Long-Term With A Specific Aldosterone Receptor Antagonist
Brief Title: Patient's Management Receiving Eplerenone Therapy
Acronym: PERGAME
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: NRA6140035
Record Dates: First submitted 2011-09-14; First posted 2011-09-26 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Left Ventricular Dysfunction Post Myocardial Infarction
Keywords: patients with MI- on top of treatment add Eplerenone - assess LVEF and BP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Eplerenone
  Interventions: Other: Prospective Observational

INTERVENTIONS:
Other: Prospective Observational — this is an observational study non interventional

SUMMARY:
On a population of patients followed by an office-based cardiologist and treated with eplerenone, the objectives of the survey are:

* To describe the characteristics of the population treated.
* To describe the methods of use of eplerenone (posology, duration of treatment, medicinal combinations).
* To describe the follow-up methods of the treatment.
* To describe the possible interruptions of the treatment

DETAILED DESCRIPTION:
A sample size in the region of N = 400 patients will allow this accuracy of estimation, as for this size, the half-width would be equal to 5% for a frequency of 50% corresponding to a confidence interval of maximum width. In view of the type of survey and the need for 12 months of monitoring in the context of standard practice, it may be anticipated that the drop-off rate will be about 20%. A sample size of N = 500 patients was therefore chosen.

ELIGIBILITY:
Inclusion Criteria:

The following patients may be selected to participate in the survey:

* Those undergoing treatment with eplerenone in accordance with the MA or not, with a known start date.
* Those likely to be followed by the same physician for a minimal period of twelve months.

Exclusion Criteria:

* Severe Kidney Disease
* Hyperkamiemia more than 5.5

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The following patients may be selected to participate in the survey:
  * Those undergoing treatment with eplerenone in accordance with the MA or not, with a known start date.
  * Those likely to be followed by the same physician for a minimal period of twelve months.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=NRA6140035&StudyName=Assessment%20Of%20Follow-Up%20Methods%20For%20Patients%20Treated%20In%20The%20Long-Term%20With%20A%20Specific%20Aldosterone%20Receptor%20Antagonist

RESULTS

PARTICIPANT FLOW:
Groups:
- Eplerenone: Participants who received eplerenone according to the approved summary of product characteristics (SmPC) were observed for 12 months. Eplerenone treatment initiated at 25 mg once daily and titrated to the target dose of 50 mg once daily within 4 weeks based on the kalaemia level.
Period: Overall Study
Arm/Group | Eplerenone
Started | 160
Completed | 155
Not Completed | 5
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Arm/Group | Eplerenone
Number analyzed (Participants) | 160
Age, Continuous [Mean (Standard Deviation); unit: Years] — Out of a total of 160 participants, data for baseline measure (age) was available for only 159 participants.
  Years | 67.70 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 121

OUTCOME MEASURES:

1. Primary Outcome: Systolic Ejection Fraction as a Measure of Left Ventricular Dysfunction at Inclusion for Full Analysis Set (FAS) Population
Description: Left ventricular dysfunction, a condition in which the left ventricle of the heart exhibits a decreased functionality, was assessed based on systolic ejection fraction. Systolic ejection fraction was the fraction of the end-diastolic volume (EDV) that was ejected out of left ventricle with each contraction.
Time Frame: Baseline
Population: FAS population included all participants who had been on study medication with inclusion questionnaire and at least one follow-up questionnaire completed, and excluded those participants with treatment start date occurring after the inclusion date. 'N' (number of participants analyzed)= participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Percentage of EDV
Arm/Group | Eplerenone
Number analyzed (Participants) | 127
Percentage of EDV | 41.2 (13.0)

2. Primary Outcome: Systolic Ejection Fraction as a Measure of Left Ventricular Dysfunction at Inclusion for Safety Analysis Set (SAS) Population
Description: as for outcome 1
Time Frame: Baseline
Population: SAS population included all participants who received study medication. Here, 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Percentage of EDV
Arm/Group | Eplerenone
Number analyzed (Participants) | 133
Percentage of EDV | 41.40 (12.82)

3. Primary Outcome: Percentage of Participants With Eplerenone Treatment Compliance at Month 3 in FAS Population
Description: Participants receiving eplerenone on the basis of the approved summary of product characteristics (SmPC) were said to be treatment compliant.
Time Frame: Month 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 90
Percentage of participants | 98.9 [94.0 to 99.8]

4. Primary Outcome: Percentage of Participants With Eplerenone Treatment Compliance at Month 6 in FAS Population
Description: Participants receiving eplerenone on the basis of the approved SmPC were said to be treatment compliant.
Time Frame: Month 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 71
Percentage of participants | 95.8 [88.3 to 98.6]

5. Primary Outcome: Percentage of Participants With Eplerenone Treatment Compliance at Month 9 in FAS Population
Description: Participants receiving eplerenone on the basis of the approved SmPC were said to be treatment compliant.
Time Frame: Month 9
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 58
Percentage of participants | 94.8 [85.9 to 98.2]

6. Primary Outcome: Percentage of Participants With Eplerenone Treatment Compliance at Month 12 in FAS Population
Description: Participants receiving eplerenone on the basis of the approved SmPC were said to be treatment compliant.
Time Frame: Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 70
Percentage of participants | 94.3 [86.2 to 97.8]

7. Primary Outcome: Percentage of Participants With Change From Baseline in Eplerenone Treatment Dosage at Month 3 in FAS Population
Description: Change of eplerenone dosage = modified dosage (mg daily) - dosage at start of treatment (mg daily). A positive change indicated dosage increase and a negative change indicated dosage decrease.
Time Frame: Baseline, Month 3
Population: FAS population. Here 'n' is signifying those participants who were evaluable for this measure at given time point for each group respectively.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 148
Percentage of participants
  Baseline: 10.7 mg daily dose (n=148) | 0.7 [0.1 to 3.7]
  Baseline: 12.5 mg daily dose (n=148) | 3.4 [1.5 to 7.7]
  Baseline: 25 mg daily dose (n=148) | 84.5 [77.8 to 89.4]
  Baseline: 50 mg daily dose (n=148) | 11.5 [7.3 to 17.6]
  Change at Month 3: Decrease (n=89) | 4.5 [1.8 to 11.0]
  Change at Month 3: No change (n=89) | 76.4 [66.6 to 84.0]
  Change at Month 3: Increase (n=89) | 19.1 [12.3 to 28.5]

8. Primary Outcome: Percentage of Participants With Change From Baseline in Eplerenone Treatment Dosage at Month 6 in FAS Population
Description: as for outcome 7
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 68
Percentage of participants
  Decrease | 5.9 [2.3 to 14.2]
  No change | 70.6 [58.9 to 80.1]
  Increase | 23.5 [15.0 to 34.9]

9. Primary Outcome: Percentage of Participants With Change From Baseline in Eplerenone Treatment Dosage at Month 9 in FAS Population
Description: as for outcome 7
Time Frame: Baseline, Month 9
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 55
Percentage of participants
  Decrease | 7.3 [2.9 to 17.3]
  No change | 60.0 [46.8 to 71.9]
  Increase | 32.7 [21.8 to 45.9]

10. Primary Outcome: Percentage of Participants With Change From Baseline in Eplerenone Treatment Dosage at Month 12 in FAS Population
Description: as for outcome 7
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 66
Percentage of participants
  Decrease | 6.1 [2.4 to 14.6]
  No change | 78.8 [67.5 to 86.9]
  Increase | 15.2 [8.4 to 25.7]

11. Primary Outcome: Percentage of Participants Who Died in SAS Population
Time Frame: Baseline up to Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 148
Percentage of participants | 6.1 [3.2 to 11.2]

12. Primary Outcome: Percentage of Participants Hospitalized in FAS Population
Time Frame: Baseline up to Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 146
Percentage of participants | 22.6 [16.6 to 30.0]

13. Primary Outcome: Number of Participants With Worsened Renal Function
Time Frame: Baseline up to Month 12
Population: Data were not analyzed because the assessment of renal function was not included in the planned analysis of this study.
Arm/Group | Eplerenone
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Participants With Reason for Increased or Decreased Eplerenone Dose
Time Frame: Baseline up to Month 12
Population: Data were not statistically summarized and were provided in individual participant listings as per the planned analysis.
Arm/Group | Eplerenone
Number analyzed (Participants) | 0

15. Secondary Outcome: Number of Participants With Concomitant Cardiovascular Treatment in FAS Population
Description: Concomitant cardiovascular treatment included any cardiovascular treatment other than, and in addition to, the study treatment taken at any time during the study.
Time Frame: Baseline up to Month 12
Population: FAS population included all participants who had been on study medication with inclusion questionnaire and at least one follow-up questionnaire completed, and excluded those participants with treatment start date occurring after the inclusion date.
Measure: Number; unit: Participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 148
Participants | 143

16. Secondary Outcome: Number of Participants With Concomitant Cardiovascular Treatment in SAS Population
Description: as for outcome 15
Time Frame: Baseline up to Month 12
Population: SAS population included all participants who received study medication.
Measure: Number; unit: Participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 160
Participants | 144

17. Secondary Outcome: Percentage of Participants Who Discontinued Eplerenone Treatment in FAS Population
Time Frame: Baseline up to Month 12
Population: FAS population. Here, 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 143
Percentage of participants | 13.3 [8.7 to 19.8]

18. Other Pre Specified Outcome: Percentage of Participants With Other Notable Events in FAS Population
Description: Other notable events included any clinically significant event other than death or hospitalization (example, ventricular tachycardia treated by defibrillator, imbalanced diabetes, work accident, right foot gout crisis, low back pain-oliguria, chest pain, bronchitis, renal failure, heart failure, hypotension, edema, standardization of gamma glutamyl transpeptidase (GT) after stopping lamisyl (peros) prescribed for a long term for mycosis, pain, nausea, fracture, trauma, gonarthrosis, increased urea, elevation of gamma GT etc.).
Time Frame: Baseline up to Month 12
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 148
Percentage of participants | 18.9 [13.4 to 26.0]

19. Other Pre Specified Outcome: Percentage of Participants With General Practitioner (GP) Consultation in FAS Population
Time Frame: Baseline up to Month 12
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 148
Percentage of participants | 77.7 [70.3 to 83.7]

20. Other Pre Specified Outcome: Number of Measurements Per Month for Kalaemia Levels in FAS Population
Description: The presence of excess potassium in the circulating blood is called hyperkalaemia. Normal potassium serum level is 3.5 to- 5.0 millimole per liter (mmol/L). Number of measurements per month for the kalaemia levels was reported.
Time Frame: Months 3, 6, 9, 12
Population: FAS population. 'N' (number of participants analyzed)= participants evaluable for this measure. Here 'n' is signifying those participants who were evaluable for this measure at given time point for each group respectively.
Measure: Mean (Standard Deviation); unit: Measurements per month
Arm/Group | Eplerenone
Number analyzed (Participants) | 92
Measurements per month
  Month 3 (n=92) | 0.5 (0.33)
  Month 6 (n=71) | 0.4 (0.27)
  Month 9 (n=58) | 0.3 (0.23)
  Month 12 (n=70) | 0.2 (0.17)

21. Other Pre Specified Outcome: Maximum Kalaemia Levels in Serum in FAS Population
Description: The presence of excess potassium in the circulating blood is called hyperkalaemia. Normal potassium serum level is 3.5 to- 5.0 mmol/L.
Time Frame: Baseline up to Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Eplerenone
Number analyzed (Participants) | 127
mmol/L | 4.6 (0.56)

22. Other Pre Specified Outcome: Change From Baseline in Maximum Value of Kalaemia Levels in FAS Population
Description: The presence of excess potassium in the circulating blood is called hyperkalaemia. Normal potassium serum level is 3.5 to- 5.0 mmol/L. Change in maximum value kalaemia level was calculated by subtracting the baseline values from the maximum observed value of kalaemia levels during the study.
Time Frame: Baseline up to Month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Eplerenone
Number analyzed (Participants) | 140
mmol/L
  Baseline (n=140) | 4.2 (0.38)
  Change in maximum Kalaemia level (n=123) | 0.4 (0.59)

23. Other Pre Specified Outcome: Percentage of Participants With Signs of Cardiac Insufficiency in FAS Population
Description: New York Health Association (NYHA) functional classification included: Class I (no limitation in physical activity, no dyspnea with normal activity), Class II (slight limitation of physical activity; fatigue, palpitation, or dyspnea with ordinary physical activity), Class III (marked limitation of physical activity; fatigue, palpitation, or dyspnea with less than ordinary physical activity) and Class IV (cannot perform a physical activity without any symptoms, dyspnea at rest). Percentage of participants in each functional class was reported.
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 148
Percentage of participants
  Baseline: Stage I (n=148) | 16.9 [11.7 to 23.7]
  Baseline: Stage II (n=148) | 54.1 [46.0 to 61.9]
  Baseline: Stage III (n=148) | 28.4 [21.7 to 36.1]
  Baseline: Stage IV (n=148) | 0.7 [0.1 to 3.7]
  Month 3: Stage I (n=91) | 29.7 [21.3 to 39.7]
  Month 3: Stage II (n=91) | 61.5 [51.3 to 70.9]
  Month 3: Stage III (n=91) | 6.6 [3.1 to 13.6]
  Month 3: Stage IV (n=91) | 2.2 [0.6 to 7.7]
  Month 6: Stage I (n=71) | 23.9 [15.5 to 35.0]
  Month 6: Stage II (n=71) | 64.8 [53.2 to 74.9]
  Month 6: Stage III (n=71) | 8.5 [3.9 to 17.2]
  Month 6: Stage IV (n=71) | 2.8 [0.8 to 9.7]
  Month 9: Stage I (n=58) | 22.4 [13.6 to 34.7]
  Month 9: Stage II (n=58) | 65.5 [52.7 to 76.4]
  Month 9: Stage III (n=58) | 12.1 [6.0 to 22.9]
  Month 12: Stage I (n=70) | 27.1 [18.1 to 38.5]
  Month 12: Stage II (n=70) | 64.3 [52.6 to 74.5]
  Month 12: Stage III (n=70) | 8.6 [4.0 to 17.5]

24. Other Pre Specified Outcome: Percentage of Participants With Reason for Starting Eplerenone Treatment in FAS Population
Description: Reasons for starting eplerenone treatment included myocardial infarction, heart failure and other conditions including severe hypertension by primary hyperaldosteronism; hypertension/coronaropathy and hypokalaemia; hypertension; left ventricular failure; not tolerated spironolactone; hypertension: gynecomastia with aldactone; pulmonary suboedema; hypertension: adrenal hyperplasia, gynecomastia with aldactone; hypertension not controlled.
Time Frame: Baseline
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eplerenone
Number analyzed (Participants) | 147
Percentage of participants
  Myocardial infarction | 61.9 [53.8 to 69.4]
  Heart failure | 29.9 [23.1 to 37.8]
  For another condition | 4.8 [2.3 to 9.5]
  Myocardial infarction and heart failure | 3.4 [1.5 to 7.7]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Eplerenone
Serious Adverse Events (participants affected / at risk) | 17/160
Other Adverse Events (participants affected / at risk) | 20/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eplerenone (N=160)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 3
Cardiac failure acute (Cardiac disorders) | 1
Cardiac flutter (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Coronary artery thrombosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal polyp (Gastrointestinal disorders) | 1
Death (General disorders) | 2
Sudden death (General disorders) | 2
Cholangitis (Hepatobiliary disorders) | 1
Erysipelas (Infections and infestations) | 1
Ejection fraction decreased (Investigations) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Coronary artery bypass (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eplerenone (N=160)
Anaemia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Condition aggravated (General disorders) | 1
Bronchitis (Infections and infestations) | 3
Ankle fracture (Injury, poisoning and procedural complications) | 1
Chest injury (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Arteriogram coronary (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Missing code (General disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 3
Gynaecomastia (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Coronary angioplasty (Surgical and medical procedures) | 1
Endarterectomy (Surgical and medical procedures) | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.